CLINICAL TRIAL: NCT03515265
Title: Clinical Performance of Direct Fiber Reinforced Resin Composite Restorations Versus Direct Microhybrid Resin Composite Restorations in Endodontically Treated Molars: A Randomized Clinical Trial
Brief Title: Clinical Performance of Fiber Reinforced Composite Versus Microhybrid Composite Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherifa Ahmed Abdelaziz Kandil, Assistant lecturer at Conservative Dentistry Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-04-22
Record Dates: First submitted 2018-04-20; First posted 2018-05-03 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: Fiber reinforced composite; Microhybrid composite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber resin composite (Experimental): Fiber reinforced resin composite restoration used as dentin substitute covered by conventional resin composite
  Interventions: Other: Fiber reinforced resin composite restoration
- Microhybrid resin composite (Active Comparator): Microhybrid resin composite restoration with lower strength compared to Fiber reinforced resin composite restoration
  Interventions: Other: Microhybrid resin composite restoration

INTERVENTIONS:
Other: Fiber reinforced resin composite restoration — a type of resin composite with improved strength due to the fiber's action
  Other Names: Ever X posterior
  Arms: Fiber resin composite
Other: Microhybrid resin composite restoration — a type of conventional resin composite
  Arms: Microhybrid resin composite

SUMMARY:
Clinical performance of direct fiber reinforced resin composite restorations versus direct microhybrid resin composite restorations in endodontically treated molars will be evaluated over 12 months using modified USPHS criteria.

DETAILED DESCRIPTION:
Restoration of endodontically treated teeth is one of the main challenges in restorative dentistry. There are structural changes in endodontically treated tooth: dehydration of dentin, mutation of collagen due to the effect of irrigation and reduction of hardness. This alteration together with loss of tooth structure inflicts a negative impact on long term prognosis of the endodontically treated tooth increases incidence of dental fracture.

Endodontically treated teeth were restored traditionally by crown but this approach is invasive with many technical and clinical steps that prolong the time of treatment. Adhesive philosophy and resin composite were developed and enhanced within the last thirty years that give clinician conservative option also strengthen, protect the tooth against fracture and changed the doctrine of devitalized tooth must be restored by crown. Current studies encourage applying conservative approach and restoring endodontically treated teeth with bonded restorations, so a lot of classic indications of crown in restoring endodontically treated teeth are questioned now.

Microhybrid resin composite restorations permit application of conservative approach that preserves remaining sound tooth structure. Fiber reinforced resin composite improved strength, toughness and fracture resistance of conventional resin composite and restored teeth.

Fiber reinforcement of conventional resin composite is introduced aiming to improve their physical, mechanical properties and tooth fracture resistance. The improvement of the properties was interpreted due to the rule of fibers in stopping crack propagation and transferring stress from matrix to fibers, also it was suggested that fiber Reinforced Resin Composites decrease polymerization shrinkage and shrinkage stress. fiber-reinforced resin composites are used as a dentine substitute combined with conventional resin composites as an enamel replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Good oral hygiene.
* Co-operative patients approving to participate in the study.
* Endodontically treated molar with minimum to moderate loss of tooth structure.
* Presence of antagonists

Exclusion Criteria:

* Patients with advanced periodontal disease.
* Patients with parafunctional habits.
* Patients with temporomandibular joint disorders.
* Teeth with failed endodontic therapy or extensive caries.
* Pregnant female

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change in the Clinical performance | Change from the baseline at six months.
  Measured using modified USPHS criteria for clinical evaluation of restoration failure.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Farid, PHD, Study Director — Professor of Conservative Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abouelleil H, Pradelle N, Villat C, Attik N, Colon P, Grosgogeat B. Comparison of mechanical properties of a new fiber reinforced composite and bulk filling composites. Restor Dent Endod. 2015 Nov;40(4):262-70. doi: 10.5395/rde.2015.40.4.262. Epub 2015 Sep 2. PMID 26587411
- See also: Fiber reinforced resin composite — https://www.gcindiadental.com/products/composite-restoratives/everx-posterior/